CLINICAL TRIAL: NCT07353814
Title: Ventilator-based Inspiratory Muscle Training: Trigger Sensitivity Adjustment Versus Stepwise Pressure Support Reduction for Patients With Respiratory Failure
Brief Title: Ventilator-based Inspiratory Muscle Training for Patients With Respiratory Failure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud El-Sayed Abduh Ragab, Assistant Lecturer Dr., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VENTILATOR-BASED TRAINING
Record Dates: First submitted 2025-12-01; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Failure; Mechanical Ventilation Complication
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: only the investigator knows the applied training method, once randomization is happened and the patient enrolled in his specific group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Chest Physiotherapy (Placebo Comparator): twenty mechanically ventilated patients with acute respiratory failure, who will receive the routine plan of weaning and conventional chest physiotherapy from MV twice a day with a 4-6 hour gap between for 4-5 days a week till extubation.
  Interventions: Other: routine plan of weaning and Conventional Chest Physiotherapy
- Trigger Sensitivity IMT (Experimental): twenty mechanically ventilated patients with acute respiratory failure, who will receive inspiratory muscle training by gradual inspiratory flow trigger sensitivity optimization in addition to the routine plan of weaning and conventional chest physiotherapy from MV, twice a day with a 4-6 hour gap between, for 4-5 days a week till extubation.
  Interventions: Other: adjustment of parameters on mechanical ventilation device; Other: routine plan of weaning and Conventional Chest Physiotherapy
- Stepwise Pressure Support Reduction IMT (Experimental): twenty mechanically ventilated patients with acute respiratory failure, who will receive inspiratory muscle training via stepwise pressure support reduction in addition to the routine plan of weaning and conventional chest physiotherapy from MV, twice a day with a 4-6 hour gap between, for 4-5 days a week till extubation.
  Interventions: Other: adjustment of parameters on mechanical ventilation device; Other: routine plan of weaning and Conventional Chest Physiotherapy

INTERVENTIONS:
Other: adjustment of parameters on mechanical ventilation device — adjust the parameters of the mode of training on mechanical ventilation according the group of patients
  Arms: Stepwise Pressure Support Reduction IMT; Trigger Sensitivity IMT
Other: routine plan of weaning and Conventional Chest Physiotherapy — Chest Physiotherapy including: ▪ Postural Drainage ▪ Manual techniques for airway clearance (percussion, vibration, shaking) Adding to range of passive to active movements of the limbs

SUMMARY:
This study will be conducted to compare the effectiveness of progressive inspiratory flow trigger sensitivity rising versus stepwise pressure support reduction as ventilator-based inspiratory muscle training methods on weaning and extubation success in mechanically ventilated patients with respiratory failure.

DETAILED DESCRIPTION:
Acute respiratory failure (ARF) remains a leading contributor to morbidity and mortality in intensive care settings. It accounts for approximately 10% to 15% of medical ICU admissions and up to 50% to 75% of prolonged ICU stays exceeding seven days, with a reported mortality rate of around 40%. Inspiratory muscle weakness is common in mechanically ventilated patients, particularly with prolonged ventilation. Inspiratory muscle training could limit or reverse these detrimental effects and promote quicker, successful weaning. Unfortunately, especially when the weaning process started late, the significant loss of muscle strength means that between 5% and 15% of patients being weaned repeatedly fail to regain respiratory autonomy. Several strategies aim to reduce weaning duration and MV time in patients requiring prolonged ventilation, including inspiratory muscle training (IMT); however, evidence for its effectiveness remains limited and inconsistent. Alternatively, ventilator-based approaches such as trigger sensitivity optimization or gradual pressure support (PS) reduction offer valid equipment-free methods that may preserve muscle activity and enhance synchrony. Despite their potential, these strategies have not been rigorously evaluated in randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory failure patients in the ICU are receiving MV for 48 h or more in a controlled mode.
* Their ages will range from 40 to 55 years old, and both sexes will be included.
* Conscious and oriented patients with a Glasgow coma score ≥13 (≥9T).
* Alertness score with a Richmond Agitation-Sedation Scale (RASS) will be from 0 to -1.
* All patients in this study must be hemodynamically and medically stable.
* Patients must be able to trigger spontaneous breaths on the ventilator but couldn't generate maximum inspiratory pressure more than -15 mbar.

Exclusion Criteria:

* Persistent hemodynamic instability as life-threatening conditions or comorbidities interfere with and compromise weaning, like cardiac arrhythmia, pericardial effusion, congestive heart failure, or acute coronary syndrome.
* Severe breathlessness when spontaneously breathing.
* Any progressive neuromuscular disease, such as myopathy or neuropathy, that would interfere with responding to inspiratory muscle training due to inadequate training performance of the inspiratory muscle.
* Spinal cord injury.
* Skeletal pathology (scoliosis, flail chest, spinal instrumentation) that would seriously impair the movement of the chest wall and ribs.
* Patients in a coma or under heavy sedation (RASS ≤ -2) and with respiratory muscle paralysis.
* High peak airway pressure (barotrauma), high PEEP >10, or active pneumothorax.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Spontaneous breathing trial (SBT) | From initiation of the first SBT until successful extubation, up to 48 hours
  documenting the frequency (total number) of spontaneous breathing trials for each patient until successful extubation
Burn's Wean Assessment Score | baseline (Day 1, prior to intervention) and immediately before initiation of successful SBT
  Calculate the percentage of the total score to indicate the extent of improvement and the probable readiness for weaning (in %). The 26-item checklist assigns 1 point for "yes" responses, with a total score up to 26. Scores below 17 (65%) suggest insufficient readiness for weaning, while scores ≥ 17 indicate probable readiness for weaning.
Duration of MV | from randomization to successful unassisted breathing, up to 48 hours
  defined as the time from study randomization to successful unassisted breathing (in days)
weaning success rate | Within 48 hours following extubation
  absence of ventilatory support 48 hours after discontinuation of MV. Inability to tolerate or pass SBT or to be liberated from invasive ventilatory support indicates weaning failure (in %).
Extubation success rate | Within 72 hours following extubation
  defined as the proportion of subjects who did not die and were not re-intubated 48-72 hours after the scheduled extubation. The inability to sustain spontaneous breathing after removal of the endotracheal tube, requiring either reintubation or the use of NIV within this specified period, indicates extubation failure (in %).

SECONDARY OUTCOMES:
Blood Gas analysis | baseline (Day 1, prior to intervention) and within 48 hours after liberation from mechanical ventilation
  Measure the results of the arterial blood gas analysis before beginning the intervention and follow up on its progression through the study and get the final results once weaning occurs. Lower PaCO₂ during MV is independently associated with successful weaning, while higher levels are linked to weaning failure
Negative Inspiratory Force | Baseline (Day 1, prior to intervention) and immediately following completion of successful SBT
  Negative inspiratory force (cmH₂O) will be measured via the mechanical ventilator as an index of global inspiratory muscle strength, consistent with ATS/ERS recommendations for weaning assessment.
Respiratory Rate | Baseline (Day 1, prior to intervention) and immediately following completion of successful SBT
  Respiratory rate (breaths/min) will be measured from the mechanical ventilator as an indicator of respiratory load and breathing pattern
Minute Ventilation | Baseline (Day 1, prior to intervention) and immediately following completion of successful SBT
  Minute ventilation (L/min) will be measured from the mechanical ventilator.
Static Lung-Thorax Compliance | Baseline (Day 1, prior to intervention) and immediately following completion of successful SBT
  Static lung-thorax compliance (mL/cmH₂O) calculated from ventilator parameters.
Rapid Shallow Breathing Index | Baseline (Day 1, prior to intervention) and immediately following completion of successful SBT
  The Rapid Shallow Breathing Index (breaths/min/L) is calculated as respiratory rate divided by tidal volume (RSBI).
The Horowitz index (also known as the oxygenation or Carrico index) | baseline (Day 1, prior to intervention) and within 48 hours after liberation from mechanical ventilation
  The PaO₂/FiO₂ ratio is a key indicator of hypoxemia severity and pulmonary recruitment in respiratory failure. Normal values range from 400 to 500 mmHg, while values below 300 mmHg indicate pulmonary dysfunction
Integrative weaning index | baseline (Day 1, prior to intervention) and immediately before initiation of successful SBT
  It is a composite parameter that was calculated as the product of static compliance (Cst), arterial oxygen saturation, and the RR/TV "RSBI":
  IWI = Cst × SaO2/RSBI (mL/cm H2O breath/minute/L). It is a reliable and accurate tool for predicting SBT outcomes and determining readiness for spontaneous breathing as an initial weaning step. An oxygen concentration of 0.35 will be preset prior to calculation, as it influences the outcome based on the formula. A value above 25 indicates a likelihood of successful weaning.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud E Ragab, M.Sc., Principal Investigator — Kasr Al Ainy hospital, Cairo University; Nesreen G' EL-NAHAS, PhD, Study Chair — Cairo University
Locations (1):
- kasr Al Ainy Hospital, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
data is available with the corresponding author on reasonable request